CLINICAL TRIAL: NCT00308334
Title: A Double Blind Placebo Controlled Trial Examining the Effect of Domperidone on the Composition of Breast Milk
Brief Title: Effect of Domperidone on the Nutrient Composition of Preterm Mother's Breast Milk
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Nurses Foundation (CNF) (Other); Dalhousie University (Other)
Responsible Party: Marsha Campbell-Yeo, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2498
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Low Breast Milk Supply
Keywords: Domperidone; breast milk; breast milk composition; preterm infant; neonate; nutrition
MeSH Terms: conditions — Premature Birth | interventions — Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Domperidone (Experimental): Domperidone
  Interventions: Drug: Domperidone
- placeob- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo- Sugar pill

INTERVENTIONS:
Drug: Domperidone — 10 mg po TID X 14 days
  Arms: Domperidone
Drug: Placebo- Sugar pill — placebo po TID x 14 days
  Arms: placeob- Sugar pill

SUMMARY:
The purpose of this study is to evaluate the effect of domperidone (given to lactating mothers of very preterm infants) on the macronutrient composition of human milk.

DETAILED DESCRIPTION:
Domperidone, a drug that enhances upper gastric motility, is an anti-dopaminergic medication that also elevates prolactin levels. It has been shown to safely increase the milk supply of lactating women. To date, researchers have analyzed the effects of domperidone on lactating woman with respect to the quantity of their milk production, adverse effects, and drug levels in the breast milk. However, the effect of domperidone on the macronutrient composition of breast milk has not been studied and current guidelines for fortification of human milk for premature infants do not distinguish between those women using or those not using domperidone. The purpose of this study is to evaluate the effect of domperidone (given to lactating mothers of very preterm infants) on the macronutrient composition of human milk.

ELIGIBILITY:
Inclusion Criteria:

* i. Mother of an infant born less than 31 weeks gestation
* ii. Women mechanically expressing breast milk using a double collecting system
* iii. Experiencing lactation failure indicated by at least one of the following: A decreasing milk supply (by greater than 30 percent from peak volume based on maternal account) An inability to provide adequate breast milk to meet the daily nutritional intake of their infant
* iv. Women who have had little or no improvement in milk production following education/counseling with a lactation consultant/Neonatal Intensive Care nurse with respect to non-pharmacological techniques.
* v. Postpartum period equal to or greater than three weeks.

Exclusion Criteria:

* i. Participants receiving any medication known to alter the effect of domperidone (e.g.cimetidine, ranitidine, famotidine, and nizatidine) or medication that interacts with domperidone (e.g. haloperidol, lithium).
* ii. Experiencing mastitis
* iii. Having a chronic or debilitating illness.
* iv. Previous breast surgery
* v. Having a known lactose intolerance

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-10; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The protein levels from breast milk will be compared, between the two groups (taking into consideration the expected rate of decline associated with increasing postpartum days). | days 0, 4, 7, and 14

SECONDARY OUTCOMES:
The fat, carbohydrate, lactose, energy, calcium, phosphorus and sodium content of breast milk will be compared between domperidone and placebo groups. | days 0, 4, 7, and 14,
Breast milk volumes (if the infant breast feeds, volume will be estimated using pre and post feeding weights) | Daily X 14 days
Serum prolactin level | Day 0, 4 and 14
infant weights | daily X 14 days
breastfeeding rates | two weeks after treatment completion and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marsha L Campbell-Yeo, MN NNP-BC PhDc, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Campbell-Yeo ML, Allen AC, Joseph KS, Ledwidge JM, Allen VM, Dooley KC. Study protocol: a double blind placebo controlled trial examining the effect of domperidone on the composition of breast milk [NCT00308334]. BMC Pregnancy Childbirth. 2006 May 23;6:17. doi: 10.1186/1471-2393-6-17. PMID 16719919
- [Derived] Campbell-Yeo ML, Allen AC, Joseph KS, Ledwidge JM, Caddell K, Allen VM, Dooley KC. Effect of domperidone on the composition of preterm human breast milk. Pediatrics. 2010 Jan;125(1):e107-14. doi: 10.1542/peds.2008-3441. Epub 2009 Dec 14. PMID 20008425